CLINICAL TRIAL: NCT05053139
Title: A Multinational, Open-label, Randomised, Controlled Study to Investigate Efficacy and Safety of NNC0365-3769 (Mim8) in Adults and Adolescents With Haemophilia A With or Without Inhibitors
Brief Title: A Research Study Investigating Mim8 in Adults and Adolescents With Haemophilia A With or Without Inhibitors
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Novo Nordisk A/S (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: NN7769-4514; U1111-1249-4378 (Other: World Health Organization (WHO)); 2020-001048-24 (Registry Identifier: European Medicines Agency (EudraCT)); jRCT2031210643 (Registry Identifier: JAPIC)
Record Dates: First submitted 2021-09-13; First posted 2021-09-22 (Actual); Last update posted 2025-12-08 (Actual); Status verified 2025-12

CONDITIONS: Haemophilia A; Haemophilia A With Inhibitors
MeSH Terms: conditions — Hemophilia A

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (5):
- no PPX- no PPX - Mim8 PPXQW/QM (Experimental): Participants not receiving prophylaxis will not enter the run-in period. In arm 1, participants will be randomised to continue no prophylaxis (on-demand treatment with their Standard of Care products) or Mim8 once-weekly or once-monthly prophylaxis in agreement with investigators in the main part of the study (26 weeks). After the main part, participants will continue in the extension part of the study (26 weeks) in agreement with the investigator, either weekly or monthly Mim8 prophylaxis regimen.
  Interventions: Drug: NNC0365-3769 (Mim8)
- no PPX - Mim8 PPXQW - Mim8 PPXQW (Experimental): Participants not receiving prophylaxis will not enter the run-in period. In arm 2a, participants will be randomised to Mim8 once-weekly prophylaxis in the main part of the study (26 weeks). After the main part, participants will continue in the extension part of the study (26 weeks) on once-weekly Mim8 prophylaxis regimen.
  Interventions: Drug: NNC0365-3769 (Mim8)
- no PPX - Mim8 PPXQM - Mim8 PPXQM (Experimental): Participants not receiving prophylaxis will not enter the run-in period. In arm 2b, participants will be randomised to Mim8 once-monthly prophylaxis in the main part of the study (26 weeks). After the main part, participants will continue in the extension part of the study (26 weeks) on once-monthy Mim8 prophylaxis regimen.
  Interventions: Drug: NNC0365-3769 (Mim8)
- PPX - Mim8 PPXQW (Experimental): Participants on coagulation factor prophylaxis prior to enrolment will preferably continue the same product type and dosing frequency in the run-in period for at least 26 weeks before they can be randomised into the main part of the study. These participants will only be allowed to receive coagulation factor prophylaxis. In arm 3, participants will be randomised to once-weekly Mim8 prophylaxis regimen in the main part of the study (26 weeks). After the main part, participants will continue in the extension part of the study (26 weeks) on once-weekly Mim8 prophylaxis regimen.
  Interventions: Drug: NNC0365-3769 (Mim8)
- PPX- Mim8 PPXQM (Experimental): Participants on coagulation factor prophylaxis prior to enrolment will preferably continue the same product type and dosing frequency in the run-in period for at least 26 weeks before they can be randomised into the main part of the study. These participants will only be allowed to receive coagulation factor prophylaxis. In arm 4, participants will be randomised to once-monthly Mim8 prophylaxis regimen in the main part of the study (26 weeks). After the main part, participants will continue in the extension part of the study (26 weeks) on once-monthly Mim8 prophylaxis regimen.
  Interventions: Drug: NNC0365-3769 (Mim8)

INTERVENTIONS:
Drug: NNC0365-3769 (Mim8) — Mim8 will be injected into a skinfold on the stomach with a thin needle either once a week or once a month.

SUMMARY:
This study is investigating how Mim8 works compared to other medicines in people with haemophilia A, who either have inhibitors or do not have inhibitors. Mim8 is a new medicine that will be used for prevention of bleeding episodes. Mim8 works by replacing the function of the missing clotting factor VIII (FVIII).

When and how often participants will receive Mim8 is dependent on their previous treatment - but is otherwise decided by chance. Mim8 will be injected into a skinfold on the stomach with a thin needle either once a week or once a month.

The study will last 54-124 weeks (12-29 months) depending on how long participants will be followed in run-in before they start treatment and if they continue in the follow period or transfer to an open label extension study. Participants will have 12-17 clinic visits.

ELIGIBILITY:
Inclusion Criteria:

1. Informed consent obtained before any study-related activities. Study-related activities are any procedures that are carried out as part of the study, including activities to determine suitability for the study.
2. Male or female participants with diagnosis of congenital haemophilia A of any severity based on medical records.
3. Participant has been prescribed treatment with factor VIII concentrates or bypassing agent in the last 26 weeks prior to screening.
4. Age above or equal to 12 years at the time of signing informed consent.
5. Body weight greater than or equal to 30 kg.
6. Applicable to participants treated with on-demand/no prophylaxis prior to enrolment: ≥5 bleeds in the last 26 weeks prior to screening visit, for which factor VIII concentrates or bypassing agent has been prescribed.
7. Applicable to participants with FVIII activity ≥1% who are on prophylactic treatment: ≥1 bleed in the last 26 weeks prior to screening visit, for which factor VIII concentrates or bypassing agent has been prescribed.
8. Willingness and ability to comply with scheduled visits and study procedures, including the completion of diary and patient-reported outcomes questionnaires.

Exclusion Criteria:

1. Previous participation in this study. Participation is defined as signed informed consent.
2. Participation (i.e., signed informed consent) in any interventional clinical study with receipt of the last dose within 6 months (or 5 half-lives of the investigational medicinal product, whichever is shorter) before planned randomisation.
3. Exposure to non-factor haemostatic products for bleeding prophylaxis within 6 months (or 5 half-lives of the medicinal product, whichever is shorter) before planned randomisation, for participants not included in the run-in.
4. Female who is pregnant, breast-feeding or intends to become pregnant or is of child-bearing potential and not using a highly effective contraceptive method. Breast feeding is allowed only during the run-in period.
5. Any disorder, except for conditions associated with haemophilia A, which in the investigator's opinion might jeopardise participant's safety or compliance with the protocol.
6. Known or suspected hypersensitivity to trial product(s), any constituents of the product or to related products.
7. Receipt of gene therapy at any given time point.
8. Ongoing or planned immune tolerance induction (ITI) therapy.
9. Major surgery planned to take place after screening.
10. Known congenital or acquired coagulation disorders other than haemophilia A.
11. Hepatic dysfunction defined as aspartate aminotransferase (AST) and/or alanine aminotransferase (ALT) above 3 times the upper limit combined with total bilirubin above1.5 times the upper limit measured at screening.
12. Renal impairment defined as estimated Glomerular Filtration Rate (eGFR) below or equal to 30 ml/min/1.73 m^2 for serum creatinine measured at screening.
13. Previous or current thromboembolic disease or events (with the exception of previous catheter-associated thrombosis for which anti-thrombotic treatment is not currently ongoing) or risk of thromboembolic disease, as evaluated by investigator.
14. Mental incapacity, unwillingness to cooperate, or a language barrier precluding adequate understanding and cooperation.
15. Other conditions (e.g., autoimmune disease) or laboratory abnormality that may increase risk of bleeding or thrombosis as evaluated by the investigator.

Min Age: 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 281 (Actual)
Dates: Start 2021-12-02 (Actual); Primary Completion 2024-03-11 (Actual); Study Completion 2024-12-17 (Actual)

PRIMARY OUTCOMES:
Number of treated bleeds | No prophylaxis treatment (Arms 1, 2a and 2b): From randomisation (week 0) to end of main (week 26)
  Count
Number of treated bleeds | Prophylaxis treatment (Arms 3 and 4): From initiation of run-in (26-52 weeks prior to week 0) to week 0 and from randomisation (week 0) to end of main (week 26)
  Count

SECONDARY OUTCOMES:
Number of injection site reactions | All participants receiving Mim8 (Arms 2a, 2b, 3 and 4): From randomisation (week 0) to end of main (week 26)
  Count
Occurrence of anti-Mim8 antibodies | All participants receiving Mim8 (Arms 2a, 2b, 3 and 4): From randomisation (week 0) to end of extension (week 52)
  Count
Number of treated spontaneous bleeds | No prophylaxis treatment (Arms 1, 2a and 2b): From randomisation (week 0) to end of main (Week 26) Prophylaxis treatment (Arms 3 and 4): From initiation of run-in (26-52 weeks prior to week 0) to week 0 and from week 0 to end of main (week 26)
  Count
Number of treated joint bleeds | No prophylaxis treatment (Arms 1, 2a and 2b): From randomisation (week 0) to end of main (Week 26) Prophylaxis treatment (Arms 3 and 4): From initiation of run-in (26-52 weeks prior to week 0) to week 0 and from week 0 to end of main (week 26)
  Count
Number of treated traumatic bleeds | No prophylaxis treatment (Arms 1, 2a and 2b): From randomisation (week 0) to end of main (Week 26) Prophylaxis treatment (Arms 3 and 4): From initiation of run-in (26-52 weeks prior to week 0) to week 0 and from week 0 to end of main (week 26)
  Count
Number of target joint bleeds | No prophylaxis treatment (Arms 1, 2a and 2b): From randomisation (week 0) to end of main (Week 26) Prophylaxis treatment (Arms 3 and 4): From initiation of run-in (26-52 weeks prior to week 0) to week 0 and from week 0 to end of main (week 26)
  Count
Consumption of factor product per bleed treatment (number of injections) | No prophylaxis treatment (Arms 1, 2a and 2b): From randomisation (week 0) to end of main (Week 26) Prophylaxis treatment (Arms 3 and 4): From initiation of run-in (26-52 weeks prior to week 0) to week 0 and from week 0 to end of main (week 26)
  Count
Change in physical function domain of PEDS-QL (pediatric quality of life inventory) | All participants (Arms 1, 2a, 2b, 3 and 4): From randomisation (week 0) to the end of the main part (week 26)
  Score points Minimum score per question (best) = 0 Maximum score per question (worst) = 4 Total score for 13 questions: 0 (best) to 92 (worst)
Change in patient's treatment burden using the Hemo-TEM (haemophilia treatment experience measure) | All participants (Arms 1, 2a, 2b, 3 and 4): From randomisation (week 0) to the end of the main part (week 26)
  Score points
  Ranges from 0 (best) - 4 (worst) representing answers ranging:
  'Not at all difficult' - 'Extremely difficult' 'Never' - 'always' 'Not at all bothered' - 'Extremely bothered' 'Not at all interfering' - 'Extremely interfering' 'Not at all burdened' - 'Extremely burdened'
Change in patient's joint pain score using Joint Pain Rating Scale | All participants (Arms 1, 2a, 2b, 3 and 4): From randomisation (week 0) to the end of the main part (week 26)
  Score points ranges from 0 = 'not at all' (best) to 4 = 'extremely' (worst)

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Transparency (dept. 2834), Study Director — Novo Nordisk A/S
Locations (163):
- United States (34):
  - Arizona H&T Phoenix Child Hosp, Phoenix, Arizona
  - Hemophilia Treatment Center, Los Angeles, California
  - Children's Hospital Los Angeles - Endocrinology, Los Angeles, California
  - Univ of Colorado Sch of Med, Aurora, Colorado
  - Univ of Miami/SCCC, Miami, Florida
  - Arnold Palmer Hospital for Children, Orlando, Florida
  - St Joseph's Hospital Foundation, Tampa, Florida
  - Children HC Atlanta-Adv Pediat, Atlanta, Georgia
  - Augusta University, Augusta, Georgia
  - Memorial Health Univ Med Ctr, Savannah, Georgia
  - Rush University Med. Cntr, Chicago, Illinois
  - Indiana Hemophilia-Thromb Ctr, Indianapolis, Indiana
  - University of Iowa_Iowa City, Iowa City, Iowa
  - University Of Iowa, Iowa City, Iowa
  - Children's Hosp-New Orleans, New Orleans, Louisiana
  - University Of Michigan, Ann Arbor, Michigan
  - Michigan State University, East Lansing, Michigan
  - Washington University School of Medicine_St. Louis, St Louis, Missouri
  - Univ of NE Med Center_Omaha, Omaha, Nebraska
  - Cure 4 the Kids Foundation, Las Vegas, Nevada
  - Torrence Hemby Ped Hem/Onc Ctr, Charlotte, North Carolina
  - St. Jude Clinic Novant Health, Charlotte, North Carolina
  - Cincinnati Child's Hsp Med Ctr, Cincinnati, Ohio
  - Univ Hosp Cleveland Med Ctr, Cleveland, Ohio
  - Nationwide Children's Hospital, Columbus, Ohio
  - Dayton Children Hemostati Ctr, Dayton, Ohio
  - Penn State MS Hershey Med Ctr, Hershey, Pennsylvania
  - St Christopher Hosp for Child, Philadelphia, Pennsylvania
  - Balad Hlth Sys-Welmont CardCVA, Kingsport, Tennessee
  - Vanderbilt Hemostasis Thrombosis Clinic, Nashville, Tennessee
  - Children's Medical Center_Dallas, Dallas, Texas
  - Univ TX Hlth Sci Ctr Houston, Houston, Texas
  - Providence Sacred Heart Medical Center & Children's Hospital, Spokane, Washington
  - Children's Hospital of Wisconsin, Milwaukee, Wisconsin
- Austria (2):
  - Universitätsklinik für Innere Medizin V, Innsbruck
  - AKH - Klin. Abt. f. Haematologie u. Haemostaseologie, Vienna
- Belgium (3):
  - Cliniques universitaires Saint-Luc - Service Hématologie, Brussels
  - UZ Antwerpen - UZA - Kinderhemato-Oncologie, Edegem
  - UZ Leuven - Kindergeneeskunde, Leuven
- Canada (9):
  - University of Manitoba, Winnipeg, Manitoba
  - St. John Regional Hospital, Saint John, New Brunswick
  - Eastern Health Authority, St. John's, Newfoundland and Labrador
  - McMaster University Medical Center, Hamilton, Ontario
  - McMaster University, Hamilton, Ontario
  - London Health Sciences Center Ontario, London, Ontario
  - The Hospital for Sick Children, Toronto, Ontario
  - Hopital Maisonneuve Rosemont, Montreal, Quebec
  - Royal University Hospital, Saskatoon, Saskatchewan
- China (14):
  - Beijing Children's Hospital, Capital Medical University, Beijing, Beijing Municipality
  - Haemotology, Nanfang Hospital, Southern Medical University, Guangzhou, Guangdong
  - Nanfang Hospital, Southern Medical University-Haematology, Guangzhou, Guangdong
  - Tongji Hospital, Tongji Medical College of HUST-Hematology, Wuhan, Hubei
  - Tongji Hospital, Tongji Medical College of HUST, Wuhan, Hubei
  - Xiangya Hospital Central-South University, Changsha, Hunan
  - The First Affiliated Hospital of Soochow University, Suzhou, Jiangsu
  - Jinan Central Hospital, Ji'Nan, Shandong
  - Jinan Central Hospital, Jinan, Shandong
  - Chengdu Women's and Children's Central Hospital, Chengdu, Sichuan
  - Institute of Hematology and Blood Diseases Hospital, Tianjin-Hematology, Tianjin, Tianjin Municipality
  - The Second Affiliated Hospital of Kunming Medical University, Kunming, Yunnan
  - Children's Hospital, Zhejiang University School of Medicine, Hangzhou, Zhejiang
  - The Children's Hospital, Zhejiang University school of medicine, Hangzhou, Zhejiang
- Ustav Hematologie a krevni tranfuze, Prague, Czechia
- Rigshospitalet - Department of Haematology, 2081, København Ø, Denmark
- France (8):
  - Centre Hospitalier Universitaire de Bordeaux-Hopital Pellegrin, Bordeaux
  - Hospices Civils de Lyon- Hopital Louis Pradel-1, Bron
  - Hôpital Cardiologique Louis Pradel, Bron
  - Ap-Hp-Hopital de Bicetre-1, Le Kremlin-Bicêtre
  - Centre Hospitalier Universitaire de Lille-Institut Coeur Poumon, Lille
  - Centre Hospitalier Universitaire de Nantes-Hopital Hotel-Dieu, Nantes
  - Ap-Hp-Hopital Necker-1, Paris
  - Centre Hospitalier Universitaire de Rennes - Hopital Pontchaillou, Rennes
- Germany (3):
  - Vivantes Netzwerk für Gesundheit GmbH - Vivantes Klinikum im Friedrichshain, Berlin
  - Universitätsklinikum Bonn - Institut für Experimentelle Hämatologie, Bonn
  - HZRM Haemophilie-Zentrum Rhein Main GmbH, Frankfurt am Main
- India (5):
  - Nirmal Hospital Pvt. Ltd., Surat, Gujarat
  - Seth GS Medical College & KEM Hospital, Mumbai, Maharashtra
  - Christian medical college, Ludhiana, Punjab
  - CMCV, Ranipet, Tamil Nadu
  - Post Graduate Institute of Child Health, Noida, Uttar Pradesh
- Ireland (2):
  - St James's CRF, Dublin, Leinster
  - CHI Crumlin Haematology, Dublin
- Sheba MC - The Israeli National Hemophilia Center, Tel Litwinsky, Israel
- Italy (2):
  - Dipartimento di Ematologia Univ. Firenze, Florence
  - IRCCS Humanitas Research Hospital - Centro Trombosi e Malattie Emorragiche, Milan
- Japan (10):
  - Nagoya University Hospital_Blood Transfusion, Aichi
  - Hospital of the University of Occupational And Environmental Health Japan, Pediatrics, Kitakyusyu-shi, Fukuoka
  - Nanbu Medical Center & Children's Medical Center, Okinawa
  - Saitama Children's Med Centre_Hematology-Oncology, Saitama
  - Shizuoka Children's Hospital, Hematology-Oncology, Shizuoka
  - Jichi Medical University Hospital_Hematology, Tochigi
  - Jichi Medical University Hospital_Pediatrics, Tochigi
  - National Center for Child Health and Development_Hematology, Tokyo
  - Tokyo Medical Univ. Hospital_Laboratory Medicine, Tokyo
  - Ogikubo Hospital_Pediatries & Blood, Tokyo
- Latvia (2):
  - Stradini Clinic of Oncology, Riga
  - Children University Clinical Hospital, Riga
- Lithuania (3):
  - Hospital of LUHS "Kauno Klinikos", Kaunas
  - Children Oncohaematology department Children's Hospital,, Vilnius
  - Vilnius University hospital Santaros klinikos, Vilnius
- Malaysia (3):
  - Hospital Queen Elizabeth 1, Kota Kinabalu, Sabah
  - Hospital Ampang, Ampang, Selangor
  - Hospital Ampang, Selangor Darul Ehsan
- Centro Multidisciplinario Para El Desarrollo Especializado De La Investigación Clínica En Yucatán S.C.P. (CEMDEICY S.C.P.), Mérida, Mexico
- Netherlands (3):
  - Academisch Medisch Centrum, Amsterdam
  - Erasmus MC, Rotterdam
  - UMC Utrecht, Van Creveldkliniek, Utrecht
- Poland (3):
  - Szpital Uniwersytecki, Oddzial Kliniczny Hematologii, Krakow, Lesser Poland Voivodeship
  - Uniwersytecki Szpital Kliniczny im. J.Mikulicza-Radeckiego, Wroclaw, Lower Silesian Voivodeship
  - Uniwersytecki Szpital Dzieciecy, Dzial Krwiolecznictwa, Lublin
- Portugal (4):
  - Unidade Local de Saúde de Coimbra, E.P.E., Coimbra
  - Unidade Local de Saúde de Santo António, E.P.E, Porto
  - Centro Hospitalar de São João_Porto, Porto
  - ULS São João, E.P.E., Porto
- Romania (4):
  - Spitalul Clinic Municipal Filantropia Craiova, Craiova, Dolj
  - Institutul Clinic Fundeni, Bucharest
  - Institut Oncologic "Prof. Dr. Ion Chiricuta" Cluj Napoca, Cluj-Napoca
  - Spitalul Clinic Municipal de Urgenta Timisoara, Timișoara
- Russia (7):
  - Reg. State Budget Healthc. Inst. Regional Clinical Hospital, Barnaul
  - SAHI Kuzbass Hospital(former Regional clinical hospital), Kemerovo
  - Children Regional Clinical Hospital, Krasnodar
  - Morozovskaya municipal children hospital, Moscow
  - National Medical Research institution of haemotology, Moscow
  - Republican Hospital n.a. V. A. Baranov, Petrozavodsk
  - City out-patient clinic 37, City Hemophilia Centre, Saint Petersburg
- King Faisal Specialist Hospital & Research Centre, Riyadh, Riyadh, Saudi Arabia
- Serbia (2):
  - Clinical Centre of Serbia, Institute for Haematology, Belgrade
  - Clinical Centre of Vojvodina, Novi Sad
- Slovakia (5):
  - Nemocnica sv. Cyrila a Metoda, UNB,Klinika hemat. a transfuz, Bratislava
  - Unilabs Slovensko, s. r. o., Košice
  - Univerzitna Nemocnica Martin, Martin
  - Vseobecna nemocnica Rimavska Sobota, Rimavská Sobota
  - Vranovska nemocnica, a.s., Vranov nad Topľou
- South Africa (2):
  - Wits Bara Clinical Trial Site, Johannesburg, Gauteng
  - Charlotte Maxeke Johannesburg Academic Hospital, Parktown, Johannesburg, Gauteng
- South Korea (3):
  - Daejeon Eulji Medical Center, Eulji University, Daejeon
  - Severance Hospital, Yonsei University Health System, Seoul
  - Kyung Hee University Hospital at Gangdong, Seoul
- Spain (3):
  - Hospital Vall d'Hebron, Barcelona
  - Hospital Universitario La Paz, Madrid
  - Hospital Regional Universitario de Málaga, Málaga
- Switzerland (3):
  - Universitätsklinik für Hämatologie, Bern
  - Zentrum für Labormedizin, Sankt Gallen
  - Universitätsspital Zürich - Klinik für Medizinische Onkologie und Hämatologie, Zurich
- Taiwan (4):
  - Kaohsiung Medical University Chung-Ho Memorial Hospital_Dept of Pediatrics, Kaohsiung City
  - Chung Shan Medical University Hospital, Taichung
  - Taichung Veterans General Hospital, Taichung
  - National Taiwan University Hospital_Dept of Hematology, Taipei
- Turkey (Türkiye) (9):
  - Gazi University, Ankara, Beşevler/Ankara
  - Gazi Üniversitesi Hastanesi- Hematoloji, Ankara, Beşevler/Ankara
  - Istanbul University Oncology Institute, Capa-ISTANBUL, Capa-ISTANBUL
  - İstanbul Üniversitesi İstanbul Tıp Fakültesi Hastanesi- Onkoloji Enstitüsü, Capa-ISTANBUL, Capa-ISTANBUL
  - Akdeniz Üniversitesi Hastanesi- Hematoloji, Antalya, Konyaaltı/ Antalya
  - Acıbadem Adana Hastanesi-Hematoloji, Adana
  - Akdeniz Universitesi, Antalya
  - Ege Universitesi Tip Fakultesi, Bornova-IZMIR
  - Ege Üniversitesi Hastanesi- Hematoloji, Bornova-IZMIR
- Ukraine (2):
  - City Clinical Hospital #4 (Dnipro) - Haematology centre, Dnipro
  - Institute of blood pathology and transfusion medicine of NAMSU - General and haematol. surgery, Lviv
- United Kingdom (4):
  - Arthur Bloom Haemophilia Centre, Cardiff
  - Royal Free Haemophilia Comprehensive Care Centre, London
  - St Thomas' Hospital - Haemostasis and Thrombosis Centre, London
  - Oxford Haemophilia Comprehensive Care Center, Oxford

IPD SHARING:
Plan to Share IPD: Yes
According to the Novo Nordisk disclosure commitment on novonordisk-trials.com
URL: http://novonordisk-trials.com

REFERENCES:
- [Derived] Ong Clausen WH, Latendorf T, Stehr R, Ezban M, Lund J. Comparative ex vivo analysis of Mim8 in thrombin generation assays triggered by activated factor XI or tissue factor. Res Pract Thromb Haemost. 2025 Oct 10;9(7):103209. doi: 10.1016/j.rpth.2025.103209. eCollection 2025 Oct. PMID 41257207